CLINICAL TRIAL: NCT02579226
Title: A Phase I, Open-Label, Multicentre Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD2811 in Patients With Advanced Solid Tumours.
Brief Title: A Phase I Study of Safety, Tolerability, and PK of AZD2811 in Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6130C00001; REFMAL 390 (Other: SCRI Development Innovations, LLC)
Record Dates: First submitted 2015-09-08; First posted 2015-10-19 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Advanced Solid Tumours
Keywords: AZD2811; Advanced solid tumours; Small-cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — AZD2811

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Part A dose-escalation will evaluate the safety and tolerability of AZD2811 monotherapy at increasing doses in patients with advanced solid tumours. Patients will receive AZD2811 on Days 1 and 4 of a 28-day cycle or Day 1 only in cycles of either 21 or 28 days.
  Interventions: Drug: AZD2811
- Part B (Experimental): Part B will include patients with relapsed or refractory small-cell lung cancer (SCLC). Patients will receive AZD2811 monotherapy at the recommended Phase 2 dose (RP2D).
  Interventions: Drug: AZD2811

INTERVENTIONS:
Drug: AZD2811 — The study will be conducted in 2 parts, dose-escalation (A) and dose-expansion (B). All patients in both parts of the study with receive AZD2811.

SUMMARY:
This Phase I study is primarily designed to evaluate the safety and tolerability of AZD2811 at increasing doses in patients with advanced solid tumours and for whom no standard of care exists. The study will be conducted in two parts, a dose-escalation phase (Part A) and a dose expansion phase (Part B). During Part A, the dose-escalation phase, patient enrolment will proceed according to a 3+3 design where the maximum tolerated dose (MTD) or the recommended Phase II dose (RP2D) could be identified. The study will also characterize the pharmacokinetic (PK) profile of AZD2811 and will explore the potential biological activity by assessing anti-tumour activity in patients. Part B will further explore PK parameters, safety, tolerability, and preliminary anti-tumour activity of the AZD2811 RP2D as monotherapy (Group 1) in patients with relapsed/refractory SCLC.

DETAILED DESCRIPTION:
This is a first-time-in-patient (FTIP) study with the nanoparticle formulation of AZD2811 primarily designed to evaluate the safety and tolerability of AZD2811 at increasing doses in patients with advanced solid tumours and for whom no standard of care exists.

The study will be conducted in two parts: Part A dose-escalation and Part B dose-expansion. In Part A, the dose-escalation phase, patient enrolment has proceeded according to a 3+3 design in order to identify the maximum-tolerated dose (MTD) or recommended Phase 2 dose (RP2D). AZD2811 monotherapy has been administered IV to patients with advanced solid tumours on Days 1 and 4 of a 28-day cycle in 6 dose levels without any relevant toxicities in the first 5 patient cohorts. In Cohort 6 (200 mg), grade 4 asymptomatic neutropenia was observed, and a dose-limiting toxicity was observed in 1 patient of the 5 evaluable patients. In Cohort 7 AZD2811 (200 mg) was given on Day 1 only of a 28-day cycle; in Cohort 8 AZD2811 (200 mg) was given on Day 1 only of a 21-day cycle. In Cohort 9, the AZD2811 dose was escalated to 400 mg on Day 1 every 21 days.

The Safety Review Committee (SRC) will review the safety and tolerability of AZD2811 for each cohort and schedule to determine the next cohorts. The study will also characterize the pharmacokinetic (PK) profile of AZD2811 and will explore potential biological activity by assessing anti-tumour activity in patients.

Once the MTD is established, Part B the dose expansion phase will continue to explore PK parameters, safety, tolerability, and preliminary anti-tumour activity of the AZD2811 RP2D as monotherapy in 21 patients with relapsed/refractory SCLC.

ELIGIBILITY:
Inclusion Criteria:

Part A Dose Escalation:

1. Histological or cytological confirmation of a solid tumour and disease progression despite standard therapy(ies), or they must be intolerant to standard therapy(ies), or no standard therapy exists.
2. Patients must have received ≤3 prior chemotherapy regimens in the metastatic setting which may have included irinotecan.

Part B Dose Expansion:

1. Patients must have received at least 1 prior platinum-based systemic therapy but no more than 3 prior systemic regimens for relapsed and/or refractory SCLC.

Inclusion Criteria All Patients:

1. Measurable or non-measurable (but evaluable disease) according to RECIST v1.1.
2. Age ≥18
3. Adequate organ system functions, as outlined by a) absolute neutrophil count (ANC) ≥1.5 X 10^9/L, b) platelets ≥100 X 10^9/L, c) hemoglobin ≥9 g/dL, d) PT/PTT/INR ≤1.5 x upper limit of normal (ULN), e) total bilirubin ≤1.5 mg/dL, f) ALT and AST ≤3.0 times the ULN if no liver involvement or ≤5 times the ULN with liver involvement, g) creatinine ≤1.5 x ULN, OR calculated or measured creatinine clearance ≥50 mL/min, OR 24-hour measured urine creatinine clearance ≥50 mL/min
4. ECOG performance status 0-1.
5. Must provide an archived tissue sample for correlative testing, if available. If archived tissue is not available, patient will still be eligible for enrolment into the study.
6. Predicted life expectancy ≥12 weeks.
7. Females of child-bearing potential should be using adequate contraceptive measures from the time of screening until 6 months after study discontinuation, should not be breast feeding and must have a negative pregnancy test prior to start of dosing. Females of non-child-bearing potential must have evidence by the following criteria at screening: a) post-menopausal defined as aged > 50 and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments, b) documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation, c) women < 50 would be considered postmenopausal if they have been amenorrhoeic for > 12 months following cessation of all exogenous hormonal treatments, and have serum follicle-stimulating hormone and luteinizing hormone levels in the postmenopausal range.
8. Sexually active males should be willing to use barrier contraception (i.e., condoms).

Exclusion Criteria:

1. Patients who have been treated with most recent radiotherapy, immunotherapy, chemotherapy or investigational drugs within ≤21 days or 5 half-lives (whichever is shorter) from enrolment (screening), and/or who have any unresolved NCI Common Terminology Criteria of Adverse Events (CTCAE) v4.03 > Grade 1 treatment-related side effect, with the exceptions of alopecia, should not be enrolled.
2. Major surgery (excluding placement of vascular access) ≤21 days from beginning of the study drug or minor surgical procedures ≤7 days. No waiting is required following implantable port and catheter placement.
3. Previous treatment with alisertib.
4. Any of the following cardiac criteria: a) Congestive heart failure (CHF) per New York Heart Association (NYHA) classification > Class II, b) Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy, c) Unstable angina or new-onset angina, d) QTcF interval >470 ms on screening ECG.
5. Active non-infectious skin disease (including any grade rash, urticarial, dermatitis, ulceration, or psoriasis, but excluding stable plaque psoriasis from the definition of active disease).
6. Patients with diarrhoea NCI CTCAE v4.03 Grade ≥2.
7. Patient has had prescription or non-prescription drugs or other products known to be strong inhibitors/inducers of CYP3A4 which cannot be discontinued prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug.
8. Any evidence of active infection, severe or uncontrolled systemic diseases including uncontrolled hypertension, active bleeding diatheses, hepatitis B, hepatitis C and human immunodeficiency virus.
9. Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 3 weeks previously and there is no evidence of central nervous system disease progression, mild neurologic symptoms, and no requirement for chronic corticosteroid therapy.
10. Treatment with haematopoietic colony-stimulating factors (e.g., G-CSF) ≤2 weeks prior to screening visit.
11. History of hypersensitivity to active or inactive excipients (e.g., PEG) of any drug in the study or drugs with similar chemical structure or class to those being investigated in the study.
12. Lactating, breastfeeding, or positive pregnancy test for female patients of child-bearing potential.
13. Concurrent conditions that in the Investigator's opinion would jeopardize compliance with the protocol.
14. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicites (DLTs) | Patients will be followed for either 21 or 28 days in Cycle 1 to determine the incidence of Dose Limiting Toxicities (DLTs).
  Maximum Tolerated Dose (MTD) will be determined in Part A of the study by assessing the incidence of Dose Limiting Toxicities (DLTs), adverse events, and abnormal laboratory results.
  DLT is defined as:
  1. Grade 4 neutropenia for > 7 days, or febrile neutropenia.
  2. Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia with bleeding.
  3. Concurrent Grade ≥3 total bilirubin, ALT or AST or alkaline phosphatase lasting > 48 hours, or any change in liver function test results consistent with Hy's Law.
  4. Grade ≥3 non-hematologic AE except: a) Grade 3 diarrhoea controlled within 4 days with standard supportive care, b) Grade 3 elevations in ALT/AST that return to meet initial eligibility criteria within 7 days of study drug interruption.
  5. Inability to receive all doses in Cycle 1 due to treatment-related toxicity.
  6. Non-haematologic toxicity of ≥ Grade 2 (at any time during treatment) that, in the judgment of the Investigator and the Medical Monitor, is dose limiting.
The incidence of adverse events | Patients will be followed for either 21 or 28 days in Cycle 1 to determine the incidence of adverse events
  Maximum Tolerated Dose (MTD) will be determined in Part A of the study by assessing the incidence of Dose Limiting Toxicities (DLTs), adverse events, and abnormal laboratory results.
  At least 3 evaluable patients will be enrolled at each dose level (3+3 design) and will be evaluated for 21 or 28 days before escalation to the next dose level can occur. If one patient experiences a DLT, an additional 3 patients will be treated with the same dose. Therefore, a maximum of up to 6 patients may be enrolled per dose level.
The incidence of abnormal laboratory results | Patients will be followed for either 21 or 28 days in Cycle 1 to determine the incidence of abnormal laboratory results.
  Maximum Tolerated Dose (MTD) will be determined in Part A of the study by assessing the incidence of Dose Limiting Toxicities (DLTs), adverse events, and abnormal laboratory results.
  At least 3 evaluable patients will be enrolled at each dose level (3+3 design) and will be evaluated for 21 or 28 days before escalation to the next dose level can occur. If one patient experiences a DLT, an additional 3 patients will be treated with the same dose. Therefore, a maximum of up to 6 patients may be enrolled per dose level.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of encapsulated AZD2811, released AZD2811, and AZD2811 metabolites | Blood will be taken from subjects in Part A Cycle 1/Day 1: pre-dose, 1, 2, 4, 6, 8, 24, and 48 hr post dose; and Day 4: pre-dose, 1, 2, 4, 6, 8, 24, 48, 96, 336, 360, and 504 hr post dose, and Cycle 2/Day 1 pre-dose and 2 hr post dose.
  PK parameters will be derived by non-compartment analysis.
Time to maximum plasma concentration (tmax) for encapsulated AZD2811, released AZD2811, and AZD2811 metabolites. | Blood will be taken from subjects in Part A Cycle 1/Day 1: pre-dose, 1, 2, 4, 6, 8, 24, and 48 hr post dose; and Day 4: pre-dose, 1, 2, 4, 6, 8, 24, 48, 96, 336, 360, and 504 hr post dose, and Cycle 2/Day 1 pre-dose and 2 hr post dose.
  PK parameters will be derived by non-compartment analysis.
Area under the plasma concentration-time curve from zero to the last measurable concentration [AUC(0-t)] for encapsulated AZD2811, released AZD2811, and AZD2811 metabolites. | Blood will be taken from subjects in Part A Cycle 1/Day 1: pre-dose, 1, 2, 4, 6, 8, 24, and 48 hr post dose; and Day 4: pre-dose, 1, 2, 4, 6, 8, 24, 48, 96, 336, 360, and 504 hr post dose.
  PK parameters will be derived by non-compartment analysis.
Area under the plasma concentration-time curve from zero extrapolated to infinity [AUC(0-inf)] for encapsulated AZD2811, released AZD2811, and AZD2811 metabolites. | Blood will be taken from subjects in Part A Cycle 1/Day 1: pre-dose, 1, 2, 4, 6, 8, 24, and 48 hr post dose; and Day 4: pre-dose, 1, 2, 4, 6, 8, 24, 48, 96, 336, 360, and 504 hr post dose.
  PK parameters will be derived by non-compartment analysis.
Terminal rate constant (λz) for encapsulated AZD2811, released AZD2811, and AZD2811 metabolites. | Blood will be taken from subjects in Part A Cycle 1/Day 1: pre-dose, 1, 2, 4, 6, 8, 24, and 48 hr post dose; and Day 4: pre-dose, 1, 2, 4, 6, 8, 24, 48, 96, 336, 360, and 504 hr post dose.
  PK parameters will be derived by non-compartment analysis.
Terminal elimination half-life for encapsulated AZD2811, released AZD2811, and AZD2811 metabolites. | Blood will be taken from subjects in Part A Cycle 1/Day 1: pre-dose, 1, 2, 4, 6, 8, 24, and 48 hr post dose; and Day 4: pre-dose, 1, 2, 4, 6, 8, 24, 48, 96, 336, 360, and 504 hr post dose.
  PK parameters will be derived by non-compartment analysis.
Volume of distribution (Vz) for encapsulated AZD2811, released AZD2811, and AZD2811 metabolites. | Blood will be taken from subjects in Part A Cycle 1/Day 1: pre-dose, 1, 2, 4, 6, 8, 24, and 48 hr post dose; and Day 4: pre-dose, 1, 2, 4, 6, 8, 24, 48, 96, 336, 360, and 504 hr post dose.
  PK parameters will be derived by non-compartment analysis.
Objective Response Rate (ORR), including the number of complete and partial responses | Patients will be assessed after every two treatment cycles (6 or 8 weeks) for up to 1 year and every 12 weeks thereafter
  Baseline tumour imaging studies [computerized tomography (CT)] scan of the chest and abdomen/pelvis) will be performed within 28 days prior to the first dose of study drug (AZD2811) and will be repeated at the completion of Cycle 2 (Week 6 or Week 8) according the RECIST v1.1.
The incidence of Stable Disease (SD) | Patients will be assessed after every two treatment cycles (6 or 8 weeks) for up to 1 year and every 12 weeks thereafter
  Baseline tumour imaging studies [computerized tomography (CT)] scan of the chest and abdomen/pelvis) will be performed within 28 days prior to the first dose of study drug (AZD2811) and will be repeated at the completion of Cycle 2 (Week 6 or Week 8) according the RECIST v1.1.
The incidence of Progressive Disease (PD) | Patients will be assessed after every two treatment cycles (6 or 8 weeks) for up to 1 year and every 12 weeks thereafter
  Baseline tumour imaging studies [computerized tomography (CT)] scan of the chest and abdomen/pelvis) will be performed within 28 days prior to the first dose of study drug (AZD2811) and will be repeated at the completion of Cycle 2 (Week 6 or Week 8) according the RECIST v1.1.
The proportion of patients surviving at 6 months will assessed in Part B. | Survival will be determined at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Burris, III, M.D., Principal Investigator — SCRI Development Innovations, LLC
Locations (6):
- United States (6):
  - Research Site, Denver, Colorado
  - Research Site, Sarasota, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Johnson ML, Wang JS, Falchook G, Greenlees C, Jones S, Strickland D, Fabbri G, Kennedy C, Elizabeth Pease J, Sainsbury L, MacDonald A, Schalkwijk S, Szekeres P, Cosaert J, Burris H 3rd. Safety, tolerability, and pharmacokinetics of Aurora kinase B inhibitor AZD2811: a phase 1 dose-finding study in patients with advanced solid tumours. Br J Cancer. 2023 May;128(10):1906-1915. doi: 10.1038/s41416-023-02185-2. Epub 2023 Mar 4. PMID 36871042